CLINICAL TRIAL: NCT03775824
Title: Faecal Analyses in Rheumatoid Arthritis Therapy: An Prospective Observational Study of the Intestinal Microbiome in Patients With Rheumatoid Arthritis Receiving Immunosuppressive Therapy
Brief Title: Faecal Analyses in Rheumatoid Arthritis Therapy
Acronym: FART
Status: Completed | Type: Observational
Sponsor: Region Skane (Other)
Responsible Party: Principal Investigator, Kristofer Andreasson, MD, PhD, Region Skane
Other Study IDs: FART1
Record Dates: First submitted 2018-12-11; First posted 2018-12-14 (Actual); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: Rheumatoid Arthritis
Keywords: microbiome; methotrexate; tnf-inhibitor; dysbiosis
MeSH Terms: conditions — Arthritis, Rheumatoid; Dysbiosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Faecal and blood samples from study participants are stored in a biorepository.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- MTX start: Patients with active rheumatoid arthritis who are either naive to methotrexate, or have not used this medicine in the last year and who are about to start therapy with methotrexate i.v. or s.c.
  Interventions: Drug: MTX start
- TNF start: Patients with active rheumatoid arthritis who are either naive to TNF-inhibitors, or have not used this medicine in the last year and who are about to start therapy with any of the following (biosimilars included); infliximab, adalimumab, etanercept, certolizumab or golimumab
  Interventions: Drug: TNF start

INTERVENTIONS:
Drug: MTX start — Patient prescribed MTX s.c. or p.o. because of active rheumatoid arthritis
  Other Names: MTX
  Groups: MTX start
Drug: TNF start — Patient prescribed TNF-inhibitor because of active rheumatoid arthritis
  Other Names: TNF
  Groups: TNF start

SUMMARY:
This study evaluates the intestinal microbiome and disease activity in patients with rheumatoid arthritis receiving immunosuppressive therapy. Patients will be analysed at two time points in reference to two predefined primary endpoints:

* Changes in intestinal microbiome
* Response to therapy

The investigators want to evaluate if successful treatment of rheumatoid arthritis coincide with specific changes in the gut flora.

DETAILED DESCRIPTION:
Methotrexate (MTX) and tumor necrosis factor (TNF) -inhibitors are two efficient medications for the treatment of rheumatoid arthritis. In a substantial number of cases however, these medications remain ineffective. At present, the scientific community has limited understanding of why some patients are resistant to these medications. The purpose of this study is to understand if the gut flora may associate with treatment response.

Recent studies have associated rheumatoid arthritis with intestinal dysbiosis. Specifically, the bacteria Prevotella copri, has been associated with this disease, an observation that has been supported also by mechanistic studies. In patients receiving methotrexate, normalization of dysbiosis has been associated with successful treatment.

This study is of observational character and integrated in the routine clinical care of patients with rheumatoid arthritis at the Rheumatology Clinic, Skane University Hospital, Lund, Sweden. Study participants are asked to deliver blood and fecal sampling at two time-points together with clinical evaluation of disease activity. With an estimated inclusion of 50 patients, at least 20 responders and 20 non-responders are expected to be included and to be compared to each other.

If successful treatment response in rheumatoid arthritis is associated with specific alterations of the gut flora, these results may guide future studies on the impact of dysbiosis and probiotics on this disease.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid arthritis according to the 2010 classification criteria
* About to start methotrexate or TNF-inhibitor because of active disease

Exclusion Criteria:

* Failure to understand protocol
* A history of alcohol abuse
* Concomitant inflammatory bowel disease
* Any history of diverticulitis
* A history of failure to comply with prescribed medication
* Ongoing biological therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study encompasses consecutive patients with rheumatoid arthritis who by their physician at the Rheumatology Clinic, Skåne University Hospital, have been prescribed any of the predefined drugs.
  Patients who are willing to comply with the study protocoll are included.
  The study population is consequently not a sample, but encompasses a majority of patients being prescribed theses medications at our University clinic.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-08-01 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Intestinal gut flora in rheumatoid arthritis | Analysis made at study start/baseline
  Intestinal gut flora based on DNA-based microbial analysis of fecal samples
Change in gut flora | Change from baseline Dysbiosis Index Score at 6 months
  Change in Dysbiosis Index Score at follow up compared to baseline.
  The Dysbiosis Index Score measures degree of intestinal dysbiosis on a scale from 1 to 5, where 5 indicates dysbiosis. The Index has been extensively described at https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5029765/
Change in disease activity/treatment response at follow up | Change from baseline DAS-28 at 6 months
  Change in Disease Activity Score 28 (DAS-28), an established index of disease activity in rheumatoid arthritis between 0-10, where 10 equals maximum activity.

SECONDARY OUTCOMES:
Adherance to immunosuppressive therapy | Analysis made at 6 months follow up
  Is the patient still prescribed the same immunosuppressant compared to baseline?
Change in intestinal concentration Prevotella | Change from baseline concentration at 6 months
  Alterations in intestinal concentrations of Prevotella bacteria according to polymerase chain reaction (PCR)-based analysis
Change in intestinal concentration Lactobacillus | Change from baseline concentration at 6 months
  Alterations in intestinal concentrations of Lactobacillus bacteria according to PCR-based analysis
Change in intestinal concentration Clostridia | Change from baseline concentration at 6 months
  Alterations in intestinal concentrations of Clostridia bacteria according to PCR-based analysis

CONTACTS AND LOCATIONS:
Overall Officials: Kristofer Andréasson, MD PhD, Principal Investigator — Skane University Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andreasson K, Alrawi Z, Persson A, Jonsson G, Marsal J. Intestinal dysbiosis is common in systemic sclerosis and associated with gastrointestinal and extraintestinal features of disease. Arthritis Res Ther. 2016 Nov 29;18(1):278. doi: 10.1186/s13075-016-1182-z. PMID 27894337
- [Background] Zhang X, Zhang D, Jia H, Feng Q, Wang D, Liang D, Wu X, Li J, Tang L, Li Y, Lan Z, Chen B, Li Y, Zhong H, Xie H, Jie Z, Chen W, Tang S, Xu X, Wang X, Cai X, Liu S, Xia Y, Li J, Qiao X, Al-Aama JY, Chen H, Wang L, Wu QJ, Zhang F, Zheng W, Li Y, Zhang M, Luo G, Xue W, Xiao L, Li J, Chen W, Xu X, Yin Y, Yang H, Wang J, Kristiansen K, Liu L, Li T, Huang Q, Li Y, Wang J. The oral and gut microbiomes are perturbed in rheumatoid arthritis and partly normalized after treatment. Nat Med. 2015 Aug;21(8):895-905. doi: 10.1038/nm.3914. Epub 2015 Jul 27. PMID 26214836
- [Background] Pianta A, Arvikar SL, Strle K, Drouin EE, Wang Q, Costello CE, Steere AC. Two rheumatoid arthritis-specific autoantigens correlate microbial immunity with autoimmune responses in joints. J Clin Invest. 2017 Aug 1;127(8):2946-2956. doi: 10.1172/JCI93450. Epub 2017 Jun 26. PMID 28650341